CLINICAL TRIAL: NCT04759651
Title: Sleep Disorders in Patients With Suspected Lung Cancer Before and After Thoracic Surgery: A Multicenter, Observational, Prospective Cohort Study
Brief Title: Sleep Disorders in Patients With Suspected Lung Cancer Before and After Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Collaborators: Marmara University (Other); Trakya University (Other); Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other); Yedikule Training and Research Hospital (Other); Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.482.IRB1.172
Record Dates: First submitted 2021-02-01; First posted 2021-02-18 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer
Keywords: sleep disorder; vats; lung cancer; robotics; thoracoscopy
MeSH Terms: conditions — Lung Neoplasms; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Functional Outcome of Sleep Questionnaire Turkish version (FOSQ-TR) — Sleep related quality of life questionnaire.
Other: Epworth Sleepiness Scale (ESS) — Subjective level of daytime sleepiness.
Other: Berlin Questionnaire — Evaluation of high-risk for Obstructive Sleep Apnea.
Other: Stop-Bang Questionnaire — Evaluation of high-risk Obstructive Sleep Apnea.
Other: Insomnia Questionnaire — Subjective evaluation of insomnia.
Other: Restless Leg Syndrome Questionnaire — Subjective evaluation of Restless Leg Syndrome.
Other: Zung Self-rating Depression Scale (SDS) — Subjective test for evaluation of depressive mood.
Other: Beck Anxiety Inventory — Subjective test for evaluation of anxiety.

SUMMARY:
The main aim of this study is to prospectively evaluate the occurrence of sleep disorders in patients undergoing thoracic surgery due to the preliminary diagnosis of lung cancer. Secondary aims include anxiety, depressive mood and functional outcomes before and 3 months after the intervention.

DETAILED DESCRIPTION:
Cancer surgery is one of the traumas that affect human life, starting from diagnostic procedures, along with the recovery process. Although 5-year survival in lung cancer has increased to 60%, there is a general prejudice that lung cancer has a poor prognosis. A preliminary diagnosis of a such condition has consequently a negative effect on the mood and sleep patterns of the patients, starting already from the beginning of the diagnostic procedures. In our study, we want to evaluate the occurrence of sleep disorders, anxiety, depressive mood and functional outcomes before and 3 months after the surgical intervention. This would also help us to better identify the patients in need for professional support for sleep disorders as well as psychiatric conditions, and thus, a better management of patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo lung resection with a pre-diagnosis of lung cancer
* Being literate or having the physical strength to answer questions.

Exclusion Criteria:

* The patient has a chronic disease such as dementia or treatment-resistant schizophrenia in which reality assessment is impaired.
* Patients who have received chemotherapy and / or radiotherapy due to their previous disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Functional Outcome of Sleep Questionnaire scores | 3 months
  Sleep related quality of life. Score range: 5-20 points, with higher scores indicating better functional status.
Change from baseline in Epworth Sleepiness Scale scores | 3 months
  Excessive daytime sleepiness. Score range: 0-24 points, with higher scores indicating greater daytime sleepiness. Scores ≥11 are generally considered to be abnormal, or positive for excessive daytime sleepiness.
Change from baseline in Berlin Questionnaire scores | 3 months
  High-risk Obstructive Sleep Apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.
Change from baseline in STOP-BANG questionnaire scores | 3 months
  High-risk Obstructive Sleep Apnea. Score range: 0-8 points, patients with a STOP-Bang score of 0 to 2 can be classified as low risk for moderate to severe OSA whereas those with a score of 5 to 8 can be classified as high risk for moderate to severe OSA.
  The STOP-BANG is an assessment tool used to help diagnose Obstructive Sleep Apnea
Change from baseline in Insomnia questionnaire scores | 3 months
  Insomnia questionnaire. Score range: 0-28 points, with higher scores indicating greater insomnia severity.
Change from baseline in Restless Legs Syndrome questionnaire scores | 3 months
  Restless Leg Syndrome questionnaire. Score range: 0-4 points, with higher scores indicating more severe symptoms

SECONDARY OUTCOMES:
Change from baseline in Zung Self-rating Depression Scale scores | 3 months
  Zung Self-rating Depression Scale. Score range: 0-80 points, most people with depression score between 50 and 69, while a score of 70 and above indicates severe depression.
Change from baseline in Beck Anxiety Inventory scores | 3 months
  Self-rating anxiety scale. Score range: 0-63 points, a total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe".

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including de-identified individual participant data will be made available to others within 6 months after the publication of this article, as will additional related documents (study protocol, statistical analysis plan, and informed consent form), for academic purposes (e.g., meta-analyses), upon request to the corresponding author, and with a signed data access agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the publication of the results
Access Criteria: Data collected for the study, including de-identified individual participant data will be made available to others within 6 months after the publication of this article, as will additional related documents (study protocol, statistical analysis plan, and informed consent form), for academic purposes (e.g., meta-analyses), upon request to the corresponding author (serus@ku.edu.tr), and with a signed data access agreement.